CLINICAL TRIAL: NCT03891056
Title: METABOLIC SURGERY FOR PATIENTS WITH TYPE 2 DM AND GRADE I OBESITY (BMI 30-35 kg/m2) WITH BAD METABOLIC CONTROL (HbA1c > 7,5%) PROTOCOL
Brief Title: Metabolic Surgery; Gastric Bypass vs Sleeve Gastrectomy; Efects Over Type 2 DM With Bad Metabolic Control (MSO1CT)
Acronym: MSO1CT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Doctor Peset (Other)
Responsible Party: Principal Investigator, Nuria Peris Tomás, Principal Investigator, Hospital Universitario Doctor Peset
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSO1CT
Record Dates: First submitted 2019-03-06; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus; Metabolic Surgery; Sleeve Gastrectomy; BPGY
Keywords: Diabetes Mellitus; Metabolic Surgery; BMI 30-35; BPGY; Vertical Gastrectomy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Randomization will be a simple one with Epidat 4.1. A number sequence will be carried out and it will be kept in opaque closed envelopes. The envelope will be opened the operation day and the surgery technique will be decided randomly, according to the randomization sequence.
Who Masked: Participant, Care Provider
Masking Description: The study will be blinded for patients, who will not know the surgery technique they will go on. Dieticians and Endocrinologists who will follow the patients up after the surgery neither will not know it, so differences in dietary recommendations will not appear with this masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric bypass (Active Comparator): Twenty patients will be randomly assigned to perform a laparoscopic gastric bypass.
  Interventions: Procedure: metabolic surgery
- Slevee gastrectomy (Active Comparator): Twenty patients will be randomly assigned to perform a sleeve gastrectomy
  Interventions: Procedure: metabolic surgery

INTERVENTIONS:
Procedure: metabolic surgery — The study will randomize patients into two arms, one where a laparoscopic gastric bypass will be performed and another that will perform slevee gastrectomy.

SUMMARY:
The aim of the study is to compare the efficacy of laparoscopic gastric bypass versus vertical gastrectomy for the resolution of DM in patients with BMI 30-35.

DETAILED DESCRIPTION:
Hyphotesis Laparoscopic gastric bypass is the elective technique in the face of sleeve gastrectomy to improve or heal type 2 diabetes mellitus in patientes with BMI 30-35 kg/m2.

MAIN AIM:

To compare cure rate through the improvement in glycated hemoglobin and fasting glycaemia after laparoscopic gastric bypass face to sleeve gastrectomy.

SECONDARY AIMS:

To quantify both insulin and oral hypoglycemic agents dose decrease. To measure weight loss and its maintenance during the follow-up in both techniques.

To compare postoperative complications. To compare postoperative pain. To compare follow-up complications.

Matherial and methods. Type of study: Randomized clinical trial double blind with two paralel groups.

RANDOMIZATION. Randomization will be a simple one with Epidat 4.1. A number sequence will be carried out and it will be kept in opaque closed envelopes. The envelope will be opened the operation day and the surgery technique will be decided randomly, according to the randomization sequence. The study will be blinded for patients, who will not know the surgery technique they will go on. Dieticians and Endocrinologists who will follow the patients up after the surgery neither will not know it, so differences in dietary recommendations will not appear with this masking.

Subjects of study The study will rely on patients with Diabetes Mellitus type 2 and grade I obesity with HbA1c higher than 7,5 % (BMI 30-35 kg/m2 and type 2 diabetes with bad glycemic control) detected in Endocrinology and Nutrition Department of Hospital Doctor Peset. Patients will go on bariatric surgery in General and Digestive Surgery Department of the same hospital. Patients who accomplish established inclusion criteria will be recruited until sample size is completed; a minimum 40 patients size is estimated (with a type I error of 5% and a power of 80%) and the will be randomized in two 20 people branches. Investigation will follow The World Medical Association and Declaration of Helsinki guidelines.

Definition of healing and improvement. Healing will be defined when HbA1c and fasting glycaemia levels are inside normal limits without needing oral hypoglycemic agents.

Improvement will be defined when decreasing medication doses for keeping normal fasting glycaemia and level of HbA1c under 6%.

Period of study:

The required one for fulfilling the sample. An inclusion of 40 patients in two years is expected.

Variable-gathering period The patient will be call for attending the external consultation of the Endocrinology and Nutrition Department of Hospital Doctor Peset. Each subject will carry out an initial study with nutritional status assesment, cardiovascular risk factors and comorbidities (hypertension, obstructive sleep apnea, dyslipidemia), as well as discarding secondary causes of obesity. In basal state, 2 days, 3, 6 and 12 months after the surgery, a blood test consisting of biochemical analysis, specific proteins, serum hormones, inmunological markers, full blood count and hemostasis will be made. The patient will carry out dietary intervention and follow-up in each phase of the process.

ELIGIBILITY:
Inclusion Criteria:

* Both sex patients aged between 18 and 65 years old
* Class I obesity (BMI 30-35 kg/m2) with bad metabolic control (DM-2 with HbA1c > 7,5%) and non-insulin anti-diabetic treatment failure (it is necessary >10 years of known diabetes evolution time, C-peptide≥ 1 ng/ml, no insulin treatment, at least two oral hypoglycemic agents treatment);
* Patients who accomplish the follow-up protocol designed by both Surgery and Endocrinology departments
* Informed consent signed

Exclusion Criteria:

* Patients who do not accomplish the previosly described inclusion criteria; Patient's refusal to take part in the study; Patients with symptomatology of gastroesophageal reflux disease or with upper gastrointestinal series compatible with this desease.

Previous bariatric surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Number of participans with normal glycosylated hemoglobin levels | 1 year after surgery
  Healing will be defined when HbA1c and fasting glycaemia levels are inside normal limits (Hb1Ac < 6%, FBG<100mg/dl) without needing oral hypoglycemic agents.

SECONDARY OUTCOMES:
Number of participants with partial remission or improvement of diabetes | 1 year after surgery
  Partial remission: Subdiabetic hyperglycemia (Hb1Ac 6%-6,4%, FBG 100-125mg/dl) in the absence anti diabetic medication.
  Improvement: statistically significant reduction in Hb1Ac and FBG not meeting criteria for remission or decrease in anti diabetic medication requirement (by one oral agent, or 1/2 reduction in dose)
Comparison of weight loss between the two techniques; bypass and sleeve. | 2 years after surgery
  To measure weight loss and its maintenance during the follow-up in both techniques. For this, the patients will be weighed in the postoperative period at month, 3, 6 12 months and then annually.
Evaluation of postoperative complications in patients undergoing bypass and slevee with Clavien-Dindo classification. | 1 month after surgery
  Grade I: any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions. Allowed therapeutic regimens are: drugs as antiemetics, antipyretics, analgesics, diuretics and electrolytes and physiotherapy. This grade also includes wound infections opened at the bedside.
  Grade II: Requiring pharmacological treatment with drugs other than such allowed for grade I complications. Blood transfusions and total parenteral nutritional also included.
  Grade III: Requiring surgical, endoscopic or radiological intervention. Grade IV: Life-threatening complication requiring IC/ICU management. Grade V: Death of a patient.
Comparison postoperative pain in sleeve and bypass with analogue assessment scale of postoperative pain. | 3 days postoperative
  The postoperative pain of the patients during the first three postoperative days will be evaluated with the visual analogue scale from 0 (no pain) to 10 (unbearable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General and Digestive Surgery of the Dr. Peset Hospital, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided